CLINICAL TRIAL: NCT00271583
Title: A Prospective, Randomized, Double Blind, Multicenter Study to Compare the Efficacy, Safety and Tolerance of CDB-2914 With Levonorgestrel as Emergency Contraception
Brief Title: Efficacy Trial of CDB 2914 for Emergency Contraception
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CCN002; N01-HD-9-3298
Record Dates: First submitted 2005-12-29; First posted 2006-01-02 (Estimated); Last update posted 2007-12-17 (Estimated); Status verified 2007-12

CONDITIONS: Emergency Contraception
Keywords: emergency contraception; antiprogestin
MeSH Terms: interventions — ulipristal; Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: CDB-2914
Drug: levonorgestrel

SUMMARY:
Objective: To compare the efficacy, safety and tolerance of a 50 mg dose of a new antiprogestin, CDB-2914 with a 0.75 mg bid dose of levonorgestrel as emergency contraception

Design: Multicenter, randomized, double blind Phase II study to compare a 50 mg dose of CDB-2914 to a 0.75 mg bid dose of levonorgestrel as emergency contraception

Subjects are randomized to receive a one-time treatment with either one dose of 50 mg CDB-2914 (followed 12 hours later by a placebo) or 2 doses of 0.75 mg of levonorgestrel with follow-up visits at 5-7 days after expected onset of menses and another visit at 12-14 days after expected onset of menses (if needed)

The primary aim is to evaluate the efficacy of CDB-2914 used by subjects as an emergency postcoital contraceptive in comparison to a group of subjects receiving levonorgestrel.

DETAILED DESCRIPTION:
Objective: To compare the efficacy, safety and tolerance of a 50 mg dose of a new antiprogestin, CDB-2914 with a 0.75 mg bid dose of levonorgestrel as emergency contraception

Design: Multicenter, randomized, double blind Phase II study to compare a 50 mg dose of CDB-2914 to a 0.75 mg bid dose of levonorgestrel as emergency contraception

Duration: A one-time treatment with either CDB-2914 or levonorgestrel with follow-up visits at 5-7 days after expected onset of menses and another visit at 12-14 days after expected onset of menses (if needed)

Treatment: A one-time treatment with one of the following:

* Two doses of 0.75 mg of levonorgestrel to be taken 12 hours apart
* One dose of 50 mg CDB-2914 and a second placebo dose to be taken 12 hours later

Study Sites: Multicenter study in the United States

Subjects: Women of reproductive age (at least 18 years) at risk of pregnancy within 72 hours of unprotected coitus

Sample Size: Approximately 811 women will be enrolled in each treatment group to obtain 1540 evaluable subjects

Outcome Evaluations

Primary: To evaluate the efficacy of CDB-2914 used by subjects as an emergency postcoital contraceptive in comparison to a group of subjects receiving levonorgestrel.

Secondary: To compare the tolerability (as measured by vomiting and nausea) of CDB-2914 used by subjects as an emergency postcoital contraceptive with that of a group of subjects receiving levonorgestrel.

Safety/Other: To assess the frequency and intensity of adverse events and the effects on the menstrual cycle of subjects administered CDB-2914 in comparison to subjects given levonorgestrel.

ELIGIBILITY:
Inclusion Criteria:

* Menstruating women at least 18 years old;
* Give voluntary, written informed consent, and agree to observe all study requirements;
* Request emergency contraception within 72 hours (3 days) after unprotected coitus, as defined by lack of contraceptive use, or condom breakage (including condoms lubricated with spermicide) or other barrier contraceptive method failure;
* Reports that all acts of unprotected coitus during the current cycle are within 72 hours prior to enrollment;
* Willing to abstain from further acts of unprotected intercourse during that cycle;
* History of regular menstrual cycles (mean length of 24-42 days with intra-individual variation of ±5 days);
* At least one normal menstrual cycle (2 menses) post delivery or abortion;
* If subject recently discontinued hormonal contraception, one normal menstrual cycle (2 menses) must have been completed before entry in the study
* For women with a recent history of Depo Provera use, the most recent injection must be at least 3 months before study entry and the subject must have had at least one normal menstrual cycle (2 menses);
* Available for follow-up for at least the next four weeks.

Exclusion Criteria:

* Currently pregnant (positive high-sensitivity urine pregnancy test);
* pregnant or breast-feeding within the past two months;
* use of hormonal methods of contraception during the current or previous two cycles;
* current user of IUD;
* tubal ligation;
* partners with history of vasectomy;
* unsure about the date of the last menstrual period (+3 days);
* irregular menstrual cycles as defined in the inclusion criteria;
* nausea and vomiting within the previous two weeks;
* impaired hypothalamic-pituitary-adrenal reserve or oral glucocorticoid replacement therapy in the last year.

Subjects cannot be currently enrolled in any other investigational trial or re-enrolled in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1672 (Actual)
Dates: Start 1999-09; Study Completion 2001-09 (Actual)

PRIMARY OUTCOMES:
Pregnancy (efficacy) | until follow-up about one week after next menses

SECONDARY OUTCOMES:
Tolerability (side effects) | until follow-up about one week after next menses
Menstrual cycle effects | until follow-up about one week after next menses

CONTACTS AND LOCATIONS:
Overall Officials: Diana Blithe, PhD, Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (6):
- United States (6):
  - California Family Health Council, Los Angeles, California
  - University of Colorado, Denver, Colorado
  - New York University, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Eastern Virginia Medical School, Norfolk, Virginia

REFERENCES:
- [Result] Creinin MD, Schlaff W, Archer DF, Wan L, Frezieres R, Thomas M, Rosenberg M, Higgins J. Progesterone receptor modulator for emergency contraception: a randomized controlled trial. Obstet Gynecol. 2006 Nov;108(5):1089-97. doi: 10.1097/01.AOG.0000239440.02284.45. PMID 17077229